CLINICAL TRIAL: NCT06716645
Title: A Real-World Evidence Study Evaluating Quality of Life Parameters Following Treatment With Robitussin
Brief Title: A Clinical Evidence Study Evaluating Quality of Life Parameters Following Treatment With Robitussin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 300233
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Common Cold; Cough
MeSH Terms: conditions — Common Cold; Cough

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robitussin Cough Syrup (Daytime) (Experimental): Participants will be instructed to take up to 20 milliliters (ml) of Robitussin Maximum Strength Cough and Chest Congestion DM syrup orally (not to exceed 6 doses in any 24-hour period) for up to 8 days or until resolution of symptoms, whichever occurs first.
  Interventions: Drug: Robitussin Maximum Strength Cough and Chest Congestion DM
- Robitussin Cough Syrup (Daytime) + Robitussin Cough Syrup (Nighttime) (Experimental): Participants will be instructed to take up to 20 ml of Robitussin Maximum Strength Cough and Chest Congestion DM syrup and up to 20 ml of Robitussin Maximum Strength Nighttime Cough DM syrup orally (not to exceed 4 doses of daytime + 1 dose of nighttime or 3 doses of daytime + 2 doses of nighttime in any 24-hour period) for up to 8 days or until resolution of symptoms, whichever occurs first.
  Interventions: Drug: Robitussin Maximum Strength Cough and Chest Congestion DM; Drug: Robitussin Maximum Strength Nighttime Cough DM

INTERVENTIONS:
Drug: Robitussin Maximum Strength Cough and Chest Congestion DM — Dextromethorphan Hydrobromide, United States Pharmacopeia (USP) 20 milligram (mg) and Guaifenesin, USP 400 mg
  Arms: Robitussin Cough Syrup (Daytime)
Drug: Robitussin Maximum Strength Cough and Chest Congestion DM — Dextromethorphan Hydrobromide, USP 20 mg and Guaifenesin, USP 400 mg
  Arms: Robitussin Cough Syrup (Daytime) + Robitussin Cough Syrup (Nighttime)
Drug: Robitussin Maximum Strength Nighttime Cough DM — Dextromethorphan Hydrobromide, USP 30 mg and Doxylamine Succinate, USP 12.5 mg
  Arms: Robitussin Cough Syrup (Daytime) + Robitussin Cough Syrup (Nighttime)

SUMMARY:
The purpose of this Real-World Evidence study is to generate real world data from participants with cough associated with the common cold, evaluating the effects in two arms with commercially available cough syrups on health-related quality of life (QoL). Arm 1 includes one cough syrup (which can be used day or night) and Arm 2 includes the daytime cough syrup and a nighttime cough syrup.

DETAILED DESCRIPTION:
This is a longitudinal, randomized, decentralized, open-label study evaluating the effect on QoL factors in participants with cough associated with the common cold in two arms using Robitussin Maximum Strength in a real-world setting. A sufficient number of adult participants (approximately 372) with symptoms of common cold will be screened for eligibility. The study expects to enroll approximately 260 eligible participants with a total of 200 participants expected to complete the study, approximately 100 in each study group. Participants will be randomized into one of two study groups (at a 1:1 ratio). Participants will be recruited through targeted advertising on social media channels and participants will not be required to physically attend any on-site visits.

ELIGIBILITY:
Inclusion Criteria:

* Participant provides a signed and dated electronic informed consent document indicating that the participant has been informed of and consents to all pertinent aspects of the study, before any assessment is performed and participant has reviewed and is willing to follow the product label.
* Participant aged 18 years or older at the time of electronic consent, inclusive of all ethnicities, races and gender identities.
* Participant reporting initiation of cough symptoms within 48 hours prior to initiation of the virtual visit.
* Participant reporting a minimum score of 5 (moderate) for cough associated with common cold symptoms and at least one other symptom of common cold (at least mild score of 3) as per the WURSS-21 symptom domains.
* Participant reporting at least one night's sleep has been disrupted in the previous 2 nights due to the symptoms of common cold.
* Participant who is willing to self-treat their cough using the study treatment.
* Participant who is in good general and mental health.
* Participant who resides in the United States (except for Hawaii and Alaska).
* Participant who owns a mobile device with access to stable internet connection and is willing to use their device to complete study surveys and assessments per the schedule of events.
* Participant who has not taken any cough products containing dextromethorphan, guaifenesin, or doxylamine (example, Robitussin, Delsym, Vicks, Mucinex), or cough drops/lozenges containing benzocaine or menthol (example, Cepacol, Halls, Ricola) or any natural cough products during the study.

Exclusion Criteria:

* Have a history of allergies (example, rash, hives, difficulty breathing, swelling of face, lips, tongue, or throat) to any medication or any kind or sensitivity to ingredients in pain, cough, cold, and flu products; including the following active ingredients found in the Research products:

  1. Active Ingredients - dextromethorphan, guaifenesin, doxylamine.
  2. Inactive Ingredients - anhydrous citric acid, carboxymethylcellulose sodium, FD&C blue no. 1, FD&C red no. 40, glycerin, liquid glucose, menthol, natural and artificial flavors, polyethylene glycol, propylene glycol, purified water, sodium benzoate, sodium citrate, sucralose, triacetin, xanthan gum.
* Participant who is currently taking medications that may interact with the study products.
* Participant who is pregnant, lactating, or plans to be pregnant or lactating during the course of the study (self-report).
* Participant who has taken any cough products containing dextromethorphan, guaifenesin, or doxylamine (example, Robitussin, Delsym, Vicks, Mucinex), or cough drops/lozenges containing benzocaine or menthol (example, Cepacol, Halls, Ricola) or any natural cough products within 7 days prior to the virtual visit.
* Have previously been diagnosed with:

  1. prostate gland enlargement or difficulty urinating.
  2. glaucoma (excessive pressure inside your eyes).
  3. asthma, chronic bronchitis, chronic cough or chronic lung disease (difficulty in breathing and cough that won't go away).
  4. Pneumonia (within the last 6 months).
  5. Coronavirus disease (COVID-19) (within the last month).
* Are taking medication(s) to treat - psychiatric / mental health conditions (example, anxiety, depression) or Parkinson's disease. Medications such as:

  1. Monoamine oxidase inhibitor (MAOI) [example, Azilect, Emsam, Marplan, Nardil] or have stopped them within the last 2 weeks per their doctor's advice.
* Are currently taking sedatives or tranquilizers (example, Ambien, Xanax, Klonopin).
* Are taking drugs for heart problems such as quinidine, amiodarone or metoprolol, antidepressants such as fluoxetine and paroxetine, or antipsychotics such as haloperidol and thioridazine.
* Participant who is currently experiencing:

  1. cough accompanied by fever, rash, or persistent headache OR
  2. cough with too much phlegm.
* Participant who is an employee of Lindus Health, either directly involved in the conduct of the study or a member of their immediate family; or a Haleon employee directly involved in the conduct of the study or a member of their immediate family.
* Participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days prior to study entry.
* Participant who has previously been enrolled in this study.
* Participant sharing the same address as another participant who has been enrolled in this study.
* Participant who, in the opinion of the investigator or delegate, should not participate in the study, including a participant who meets any of the "stop use" criteria recommended by the label.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2024-12-04 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Wisconsin Upper Respiratory Symptom Survey-21 (WURSS-21) Total Score | Baseline and up to Day 8
  The WURSS is an evaluative illness-specific quality of life instrument, designed to assess the negative impact of acute upper respiratory infection, presumed viral (the common cold). WURSS-21 is the short version of this validated survey. Participants will rate their cold symptoms (10 questions) and QoL related 9 questions using WURSS-21. The responses will be evaluated on a scale ranging from 0 to 7, where 0=Do not have symptoms/Not at all and 7=Severe symptoms/Severely. Thus, the minimum and maximum possible total scores will be 0 and 133 respectively, where higher total scores indicate more negative impact on symptoms and quality of life. Baseline will be defined as Day 0. Change from Baseline will be calculated as each post-Baseline value minus Baseline value.
Change from Baseline in WURSS-21 Total Symptom Domain Score | Baseline and up to Day 8
  The WURSS is an evaluative illness specific quality of life instrument, designed to assess the negative impact of acute upper respiratory infection, presumed viral (the common cold). WURSS-21 is the short version of this validated survey. The symptom domain of WURSS-21 consists of 10 questions. Participants will rate their cold symptoms related questions and the responses will be evaluated on a scale ranging from 0 to 7, where 0=Do not have symptoms and 7=Severe. Thus, the minimum and maximum possible total score will be 0 and 70 respectively, where higher scores indicate more negative impact on symptoms. Baseline will be defined as Day 0. Change from Baseline will be calculated as each post-Baseline value minus Baseline value.
Change from Baseline in WURSS-21 Total QoL Domain Score | Baseline and up to Day 8
  The WURSS is an evaluative illness specific quality of life instrument, designed to assess the negative impact of acute upper respiratory infection, presumed viral (the common cold). WURSS-21 is the short version of this validated survey. The QoL domain of WURSS-21 consists of 9 questions. Participants will rate their QoL related questions and the responses will be evaluated on a scale ranging from 0 to 7, where 0=Not at all and 7=Severely. Thus, the minimum and maximum possible total scores will be 0 and 63 respectively, where higher scores indicate more negative impact on QoL. Baseline will be defined as Day 0. Change from Baseline will be calculated as each post-Baseline value minus Baseline value.
Change from Baseline in Each of the WURSS-21 Symptom Scores (10 Items in Total) | Baseline and up to Day 8
  The WURSS is an evaluative illness specific quality of life instrument, designed to assess the negative impact of acute upper respiratory infection, presumed viral (the common cold). WURSS-21 is the short version of this validated survey. The individual symptoms include runny nose, plugged nose, sneezing, sore throat, scratchy throat, cough, hoarseness, head congestion, chest congestion and feeling tired. Participants will rate each of the 10 individual symptom domain questions and the responses will be evaluated on a scale ranging from 0 to 7, where 0=Do not have symptom and 7=Severe. Thus, the minimum and maximum score for each symptom domain question will be 0 and 7, where higher scores indicate more negative impact on symptoms. Baseline will be defined as Day 0. Change from Baseline will be calculated as each post-Baseline value minus Baseline value.
Change from Baseline in Each of the WURSS-21 QoL Questions Scores (9 Items in Total) | Baseline and up to Day 8
  The WURSS is an evaluative illness specific quality of life instrument, designed to assess the negative impact of acute upper respiratory infection, presumed viral (the common cold). WURSS-21 is the short version of this validated survey. The QoL domain of WURSS-21 consists of 9 questions. Participants will rate each QoL questions, and the responses will be evaluated on a scale ranging from 0 to 7, where 0=Not at all and 7=Severely. Thus, the minimum and maximum possible total scores will be 0 and 7 respectively, where higher scores indicate more negative impact on QoL. Baseline will be defined as Day 0. Change from Baseline will be calculated as each post-Baseline value minus Baseline value.

SECONDARY OUTCOMES:
Change from Baseline in QoL Factors Assessed Using Specific QoL Questions | Baseline and up to Day 8
  QoL factors will be assessed using specific questions related to social activities, feeling self-conscious around people, coughing in public, falling asleep, sleeping through the night, energy, and motivation. Participants will rate their response to questions on a scale ranging from 0 to 7, where 0= Not at all and 7= Severely. Thus, the minimum and maximum score for each question will be 0 and 7 respectively, where higher scores indicate more negative impact on QoL. Baseline will be defined as Day 0. Change from Baseline will be calculated as each post-Baseline value minus Baseline value.
Change from Baseline in Categorized QoL Questions Score: Sleep Quality | Baseline and up to Day 8
  The QoL factors will be categorized into 4 categories - Sleep quality, Vitality, Physical activity and Social activity. Sleep quality category will include 3 individual questions - Sleep well (WURSS-21: Question 13), Falling asleep (QoL: Question 4) and Sleep through the night (QoL: Question 5). Participants will rate each question and the responses will be evaluated on a scale ranging from 0 to 7, where 0=Not at all and 7=Severely. The individual question score will be added to derive categorized QoL score. Thus, the minimum and maximum possible total scores will be 0 and 21 respectively, where higher scores indicate more negative impact on QoL. Baseline will be defined as Day 0. Change from Baseline will be calculated as each post-Baseline value minus Baseline value.
Change from Baseline in Categorized QoL Questions Score: Vitality | Baseline and up to Day 8
  The QoL factors will be categorized into 4 categories - Sleep quality, Vitality, Physical activity and Social activity. Vitality category will be assessed using 3 individual questions - Energy (QoL: Question 6), Motivation (QoL: Question 7), and Feel tired (WURSS-21: Question 11). Participants will rate each question and the responses will be evaluated on a scale ranging from 0 to 7, where 0=Not at all and 7=Severely. The individual question score will be added to derive categorized QoL score. Thus, the minimum and maximum possible total scores will be 0 and 21 respectively, where higher scores indicate more negative impact on QoL. Baseline will be defined as Day 0. Change from Baseline will be calculated as each post-Baseline value minus Baseline value.
Change from Baseline in Categorized QoL Questions Score: Physical Activities | Baseline and up to Day 8
  The QoL factors will be categorized into 4 categories - Sleep quality, Vitality, Physical activity and Social activity. Physical Activities will be assessed using 3 individual questions - Breathe easily (WURSS-21: Question 14), Walk, climb stairs, exercise (WURSS-21: Question 15) and Accomplish daily activities (WURSS-21: Question 16). Participants will rate each question and the responses will be evaluated on a scale ranging from 0 to 7, where 0=Not at all and 7=Severely. The individual question score will be added to derive categorized QoL score. Thus, the minimum and maximum possible total scores will be 0 and 21 respectively, where higher scores indicate more negative impact on QoL. Baseline will be defined as Day 0. Change from Baseline will be calculated as each post-Baseline value minus Baseline value.
Change from Baseline in Categorized QoL Questions Score: Social Activities | Baseline and up to Day 8
  The QoL factors will be categorized into 4 categories - Sleep quality, Vitality, Physical activity and Social activity. Social Activities will be assessed using 4 individual questions - Interact with others (WURSS-21: Question 19), Less comfortable in social activities (QoL: Question 1), Self-conscious around others (QoL: Question 2) and Coughing in public (QoL: Question 3). Participants will rate each question and the responses will be evaluated on a scale ranging from 0 to 7, where 0=Not at all and 7=Severely. The individual question score will be added to derive categorized QoL score. Thus, the minimum and maximum possible total scores will be 0 and 28 respectively, where higher scores indicate more negative impact on QoL. Baseline will be defined as Day 0. Change from Baseline will be calculated as each post-Baseline value minus Baseline value.

CONTACTS AND LOCATIONS:
Locations (1):
- Lindus Health Limited, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.